CLINICAL TRIAL: NCT02076373
Title: Erythropoietin for the Repair of Cerebral Injury in Very Preterm Infants - a Randomized, Double-blind, Placebo-controlled, Prospective, and Multicenter Clinical Study
Brief Title: Erythropoietin for the Repair of Cerebral Injury in Very Preterm Infants
Acronym: EpoRepair
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EpoRepair; 2013DR3204 (Other: Swissmedic)
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Intraventricular Hemorrhage of Prematurity
MeSH Terms: interventions — epoetin beta; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- recombinant human Erythropoietin (Epo) (Experimental): Epo 2000 U in normal saline per ml/kg of body weight 5 times intravenously, total dosage 10000 U per 5ml/kg.
  In detail: For loading 3 times beginning at day 5 of life (± 2 days), followed at 24 hours and 48 hours later. For maintenance 2 times, at day 10 and day 17 after the first study medication.
  Interventions: Drug: recombinant human Erythropoietin
- Control (Placebo Comparator): Placebo 1 ml normal saline/kg of body weight 5 times intravenously, total dosage 5 ml/kg.
  In detail: For loading 3 times beginning at day 5 of life (± 2 days), followed at 24 hours and 48 hours later. For maintenance 2 times, at day 10 and day 17 after the first study medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: recombinant human Erythropoietin — i.v. administration
  Other Names: Epoetin beta
  Arms: recombinant human Erythropoietin (Epo)
Drug: Placebo — i.v. administration
  Other Names: normal saline
  Arms: Control

SUMMARY:
The purpose of this randomized and placebo-controlled EpoRepair trial is to evaluate the effect of intravenously administered recombinant human erythropoietin (Epo) as compared to placebo in preterm infants with brain damage on neurological development until five years od age.

DETAILED DESCRIPTION:
Worldwide, 1% of all infants are born very preterm with less than 32 weeks of gestation, which is more than 2 months before expected date of delivery. If these smallest infants suffer in addition to prematurity a second hit, such as intraventricular hemorrhage or parenchymal infarction, they are at high risk for learning disabilities, mental retardation, and cerebral palsy in later life.

Intraventricular hemorrhage and parenchymal infarction occur in about 12% of very preterm infants, mostly in the very smallest and within the first few days after birth, and can be recorded by cranial ultrasound. Except for shunt insertion to divert cerebrospinal fluid in infants with posthemorrhagic hydrocephalus and possibly the removal of blood clots, there is no treatment for established intracerebral bleeding, and no medical therapies exist to ameliorate the neurodevelopmental sequelae.

Apart from stimulating production of red blood cells in the bone marrow, recombinant human erythropoietin (Epo) has been shown to exert neuroprotective action in a variety of animal models and in clinical studies. Epo administration has been found to be beneficial and safe in randomized controlled trials (RCT) involving adult and infant patients.

Observational data suggest that Epo administered to very preterm infants in order to prevent from anemia improves long-term cognitive outcomes until school-age especially in those infants who had suffered intracerebral bleeding. These data, however, are observational and therefore do not allow for any firm conclusions or recommendations. The hypothesis generated by these data calls for confirmation or refutation by an RCT designed to address this question.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with less than 32 weeks of gestation and/or less than 1500 g weight at birth
2. Intraventricular hemorrhage and/or hemorrhagic parenchymal infarction
3. Less than 8 days of life
4. Informed written parental consent

Exclusion Criteria:

1. Genetically defined syndrome
2. Severe congenital malformation adversely affecting life expectancy and/or neurodevelopment
3. A priory palliative care
4. Unlikely to participate at 5-year follow-up examination

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | 5 years
  With 5 years of age, composite intelligence quotient to be assessed by standardized IQ tests.

SECONDARY OUTCOMES:
Biomarker cranial MRI | 40 weeks postmenstrual age
  Brain injury score assessed on cranial MRI, including brain maturation score and white matter and gray matter injury scores, as biomarker for long-term neurodevelopmental outcome.
Safety | Infants will be followed for the duration of hospital stay, an expected average of 14 weeks
  Analysis will be performed to get insight about the distributions of adverse events and other safety relevant outcomes between groups.
Neurodevelopmental outcome | 2 years
  Bayley Scales of Infant Development (BSID-III) and the presence or absence of impairment of motor function (cerebral palsy) and neurosensory function (blindness or deafness) will be assessed with 18 to 24 months.
Biomarker serial cranial ultrasound | Infants will be followed for the duration of hospital stay, an expected average of 14 weeks
  Cranial ultrasound is a useful point of care method to detect, confirm and monitor brain damage including intracerebral bleeding. It is part of clinical routine for the duration of hospital stay.
Overall developmental outcome | 5 years
  Neurological and formal psychological examination. Normal Overall developmental outcome is classified as normal if IQ >84 and without one or more of the following: motor impairment, cognitive impairment, behavior problems, poor general health, severe hearing loss, or bilateral blindness.

OTHER OUTCOMES:
Course of intracerebral bleeding | Infants will be followed for the duration of hospital stay, an expected average of 14 weeks
  Course of intracerebral bleeding from onset until term equivalent age with additional visits at 28 days of life and 36 weeks postmenstrual age.
  1. No remaining lesions as recorded by cranial ultrasound
  2. Persisting posthemorrhagic hydrocephalus without any drainage
  3. Persisting posthemorrhagic hydrocephalus with repetitive but transient csf-drainage
  4. Posthemorrhagic hydrocephalus with permanent csf-drainage
  5. Convulsions and other abnormalities or medications related to intracerebral bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Sven Wellmann, MD, Principal Investigator — University of Zurich; Hans Ulrich Bucher, MD, PhD, Study Chair — University of Zurich
Locations (8):
- Medical University of Vienna, Vienna, Austria
- Switzerland (7):
  - Kantonsspital Aarau, Aarau
  - University Children's Hospital Basel (UKBB), Basel
  - University Hospital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruegger CM, Hagmann CF, Buhrer C, Held L, Bucher HU, Wellmann S; EpoRepair Investigators. Erythropoietin for the Repair of Cerebral Injury in Very Preterm Infants (EpoRepair). Neonatology. 2015;108(3):198-204. doi: 10.1159/000437248. Epub 2015 Aug 8. PMID 26278911
- [Derived] Wellmann S, Hagmann CF, von Felten S, Held L, Klebermass-Schrehof K, Truttmann AC, Knopfli C, Fauchere JC, Buhrer C, Bucher HU, Ruegger CM; Erythropoietin for the Repair of Cerebral Injury in Very Preterm Infants (EpoRepair) Investigators. Safety and Short-term Outcomes of High-Dose Erythropoietin in Preterm Infants With Intraventricular Hemorrhage: The EpoRepair Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244744. doi: 10.1001/jamanetworkopen.2022.44744. PMID 36459138
- See also: EpoRepair trial homepage — http://www.eporepair.ch